CLINICAL TRIAL: NCT02073500
Title: Prospective Observational Study of Peritoneal Surface Malignancies (PSM) - Characterization, Models and Treatment Strategies.
Brief Title: Peritoneal Surface Malignancies - Characterization, Models and Treatment Strategies
Acronym: PSM
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Kjersti Flatmark, Professor, Oslo University Hospital
Other Study IDs: PSM_250913
Record Dates: First submitted 2014-02-17; First posted 2014-02-27 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Pseudomyxoma Peritonei; Colorectal Carcinoma; Ovarian Carcinoma; Mesothelioma
Keywords: Peritoneal carcinomatosis; Peritoneal surface malignancy; Cytoreductive surgery; Hyperthermic intraperitoneal chemotherapy; CRS; HIPEC; Prognostic biomarker; Predictive biomarker
MeSH Terms: conditions — Pseudomyxoma Peritonei; Colorectal Neoplasms; Ovarian Neoplasms; Mesothelioma; Peritoneal Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Metastatic tissue, blood specimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational study: Patients diagnosed with PSM undergoing CRS with HIPEC.
  Interventions: Other: Observational study.

INTERVENTIONS:
Other: Observational study. — Analysis of metastatic tissue and blood specimens collected from patients with PSM undergoing CRS-HIPEC. CRS: Removal of all macroscopically detectable tumor.
  HIPEC: Instillation of heated chemotherapy in the abdominal cavity to remove residual cancer disease.
  Other Names: Observational study. Laboratory biomarker analysis.

SUMMARY:
The aim of this study is to identify biomarkers of disease recurrence and prognosis to optimize patient selection for treatment with cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC), and through animal models to explore different treatment strategies for peritoneal surface malignancies (PSM).

DETAILED DESCRIPTION:
The handling of patients with PSM involves multimodal and multidisciplinary treatment strategies such as CRS, the removal of all macroscopically detectable tumor, and HIPEC, instillation of heated chemotherapy in the abdominal cavity to remove residual cancer disease. The treatment is challenging and complex and associated with significant morbidity. Only patients with limited disease will benefit from the treatment, and better methods for patient selection are needed. The project group has a unique opportunity to address key questions because of acquired experience, an exceptional biobank and institutional database and novel animal models established at the Norwegian Radium Hospital.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* confirmed diagnosis of peritoneal surface malignancy
* candidate for CRS-HIPEC
* written informed consent

Exclusion Criteria:

* none

Approximately 80 patients per year will be eligible for inclusion, as this is the number of patients that annually receive surgical treatment for PSM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with PSM that are referred to Oslo University Hospital and are candidates for CRS with HIPEC may be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-09 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  Time from surgery until death from any cause

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  Time from surgery until disease recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Flatmark, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- The Norwegian Radium Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lund-Andersen C, Nakken S, Nygard S, Fromm B, Aasheim LB, Davidson B, Julsrud L, Abrahamsen TW, Kristensen AT, Dybdahl B, Larsen SG, Hovig E, Flatmark K. Integrative genomic analysis of peritoneal malignant mesothelioma: understanding a case with extraordinary chemotherapy response. Cold Spring Harb Mol Case Stud. 2019 Apr 1;5(2):a003566. doi: 10.1101/mcs.a003566. Print 2019 Apr. PMID 30862609